CLINICAL TRIAL: NCT05409911
Title: A Phase 1, Open-label, Parallel-group Study to Assess the Pharmacokinetics, Safety, and Tolerability of S-217622 in Participants With Mild and Moderate Hepatic Impairment and Healthy Control Participants
Brief Title: A Study to Assess S-217622 in Participants With Mild and Moderate Hepatic Impairment and Healthy Control Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2127T1213
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — ensitrelvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- S-217622: Group A (Experimental): Participants with mild hepatic impairment will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622
- S-217622: Group B (Experimental): Participants with moderate hepatic impairment will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622
- S-217622: Group C (Experimental): Participants with normal hepatic function will receive a single dose of S-217622 on Day 1, in a fasted state.
  Interventions: Drug: S-217622

INTERVENTIONS:
Drug: S-217622 — Tablet for oral administration

SUMMARY:
The objective of this study is to assess the pharmacokinetics (PK), safety, and tolerability of S-217622 in participants with mild and moderate hepatic impairment compared with control participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥50 kilograms (kg) and body mass index (BMI) within the range of ≥18.5 to <38.0 kilogram-meter squared (kg/m^2) at the Screening visit.

Participants With Hepatic Impairment

* A diagnosis of clinically stable hepatic disease for at least 1 month prior to the Screening visit, confirmed by medical history or previous confirmation of hepatic cirrhosis by liver biopsy or medical imaging technique (including laparoscopy, computerized tomography [CT] scan, magnetic resonance imaging [MRI], or ultrasonography).
* Mild or moderate hepatic impairment based on the Child-Pugh classification score at the Screening visit to determine eligibility:

  1. Mild (Class A) hepatic impairment (Child-Pugh classification score 5 to 6)
  2. Moderate (Class B) hepatic impairment (Child-Pugh classification score 7 to 9)
* A stable medication regimen is required, defined as not starting new drug(s) or changing dosage(s) within 14 days prior to administration of study intervention through the Follow-up/Early Termination visit.

Healthy Participants

* Matched to each participant with moderate (and mild when possible) hepatic impairment with respect to sex, age (± 5 years), and BMI (± 10%).

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, renal, gastrointestinal (GI), endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* History of GI surgery including but not limited to gastric resection and/or intestinal resection that resulted in a clinically significant abnormality in GI function.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Participant with poor venous access.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Time to Maximum Plasma Concentration (Tmax) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Area Under the Plasma Concentration-Time Curve (AUC) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Terminal Elimination Half-Life (t1/2,z) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Terminal Elimination Rate Constant (λz) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Mean Residence Time (MRT) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Apparent Total Clearance (CL/F) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Apparent Volume of Distribution (Vz/F) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Renal Clearance (CLR) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Fraction of Dose Excreted in Urine (Feu) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15
Fraction Unbound in Plasma (FU) of S-217622 | 0 (predose) up to 336 hours postdose on Day 1 to Day 15

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events | Up to Day 21

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Orlando Clinical Research Center, Inc., Orlando, Florida
  - Nucleus Network, Saint Paul, Minnesota